CLINICAL TRIAL: NCT04896801
Title: Prospective Study of MR-guided Prostate Stereotactic Body Radiotherapy in Seven Days
Brief Title: MR-guided Prostate Stereotactic Body Radiotherapy in Seven Days
Acronym: Proseven
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Mark De Ridder, Principal Investigator, Universitair Ziekenhuis Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO7
Record Dates: First submitted 2021-05-13; First posted 2021-05-21 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Prostate Cancer
Keywords: MR-guided radiotherapy; Stereotactic body radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- MR-guided prostate stereotactic body radiotherapy (Experimental): Patients will receive MR-guided RT in 5 fractions over 7 days (daily excluding weekend, i.e. start on Wednesday or Thursday, until Tuesday or Wednesday respectively the week after).
  Interventions: Radiation: MR-guided RT

INTERVENTIONS:
Radiation: MR-guided RT — The dose to the planning target volume (PTV) is 36 Gy (5 x 7.2 Gy) prescribed on the 90% isodose line. The clinical target volume (CTV) is receiving 40 Gy (5 x 8 Gy = 100%). A simultaneous integrated boost (SIB) up to a total dose of 42 Gy (5 x 8.4 Gy = 105%) is delivered to the gross tumor volume (GTV), if present. In addition, relative sparing of the urethra will be applied by avoiding hotspots (V40 Gy < 1cc) in the urethra. Baseline and adapted treatment plans are generated using intensity-modulated RT

SUMMARY:
The Proseven trial is a prospective interventional study that will evaluate the toxicity and efficacy of MR-guided stereotactic body radiotherapy (SBRT) in the profound hypofractionated treatment of prostate cancer. Patients will be treated in 5 daily fractions within a short overall treatment time (OTT) of 7 days. A simultaneous integrated boost (SIB) will be delivered to the intraprostatic dominant lesion (if present) in this study. Besides a potential biological impact of this innovative prostate SBRT treatment, the reduced OTT offers also benefits in terms of patient convenience. The primary endpoint is clinician reported grade 2 or more acute gastrointestinal (GI) and genitourinary (GU) toxicity, assessed using CTCAE v 5.0 and RTOG, measured up to 3 months after the first treatment fraction.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 y
* Histologically confirmed prostate adenocarcinoma
* Low risk: cT1c-T2a, Gleason score 6, PSA < 10ng/mL
* Favorable intermediate risk: 1 intermediate risk factor, Gleason 3+4 or less, < 50% positive biopsy cores)
* Unfavorable intermediate risk: > 1 intermediate risk factor, Gleason 4+3, > 50% positive biopsy cores)
* Limited high risk: cT3a with PSA < 40ng/mL or cT2a-c with a Gleason score > 7 and/or a PSA > 20ng/mL but < 40ng/mL
* World Health Organization performance score 0-2
* Written informed consent

Intermediate risk factors: T2b-T2c, Gleason 7, PSA 10-20 ng/mL

Exclusion Criteria:

* Transurethral resection (TUR) < 3months before SBRT
* International Prostate Symptom Score (IPSS) > 19
* Prostate volume > 100cc on transrectal ultrasound (TRUS)
* Stage cT3b-T4
* N1 disease (clinically or pathologically)
* M1 disease (clinically or pathologically)
* PSA > 40ng/mL
* inflammatory bowel disease
* immunosuppressive medications
* prior pelvic RT
* contra-indications for MRI

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2021-08-10 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Acute toxicity according to CTCAE v 5.0 | from the first treatment fraction up to 3 months
  Clinician reported grade 2 or more acute gastrointestinal (GI) or genitourinary (GU) toxicity, assessed using CTCAE v 5.0
Acute toxicity according to RTOG criteria | from the first treatment fraction up to 3 months
  Clinician reported grade 2 or more acute gastrointestinal (GI) or genitourinary (GU) toxicity, assessed using RTOG criteria

SECONDARY OUTCOMES:
Late toxicity according to CTCAE v 5.0 | within 5 years after start of radiotherapy
  Clinician reported late toxicity, assessed using CTCAE v 5.0
Late toxicity according to RTOG criteria | within 5 years after start of radiotherapy
  Clinician reported late toxicity, assessed using RTOG criteria
Quality of life assessment | from the start of radiotherapy until 5 years after treatment
  Quality of life according to EORTC Quality of life Questionnaire C30
Prostate specific quality of life assessment | from the start of radiotherapy until 5 years after treatment
  Quality of life according to EORTC Quality of life Questionnaire PR25
EPIC-26 quality of life | from the start of radiotherapy until 5 years after treatment
  Quality of life according to Expanded Prostate Index Composite-26 (EPIC-26)
IPSS quality of life | from the start of radiotherapy until 5 years after treatment
  Quality of life according to International Prostate Symptom Score (IPSS)
Freedom from biochemical failure | from start of radiotherapy until PSA relapse, assessed up to 5 years
  the Phoenix definition is used to define PSA failure (i.e. nadir + 2ng/mL)
Disease-free survival | from start of radiotherapy until 5 years after treatment
  from start of radiotherapy until first evidence of recurrence (loco-regional or distant) or death from any cause
Overall survival | from start of radiotherapy until 5 years after treatment
  from start of radiotherapy until death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Mark De Ridder, MD, Principal Investigator — Department of Radiotherapy, UZ Brussel, Vrije Universiteit Brussel
Locations (1):
- Department of Radiotherapy, UZ Brussel, Vrije Universiteit Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No